CLINICAL TRIAL: NCT06522620
Title: Posterior Femoral Cutaneous Nerve Combined With Proximal Sciatic and Saphenous Nerve Block for Postoperative Posterior Lateral Knee Analgesia in Patients With TKA: a Single-center, Prospective, Randomized Controlled Study
Brief Title: Effect of Posterior Femoral Cutaneous Nerve Block on Postoperative Posterior Lateral Knee Analgesia in Patients With TKA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: General Hospital of Ningxia Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Peng Liu-2024-1
Record Dates: First submitted 2024-07-16; First posted 2024-07-26 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-07

CONDITIONS: Postoperative Pain
Keywords: Posterior Femoral Cutaneous Nerve; Nerve Block; TKA; posterior lateral knee pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sciatic saphenous nerve block group (Group S) (Active Comparator): Postoperative analgesia using subgluteal approach sciatic nerve block + saphenous nerve block
  Interventions: Procedure: Simple Sciatic and Saphenous Nerve Blocks
- Combined posterior femoral cutaneous nerve block group (Group P) (Experimental): Postoperative analgesia using supragluteal approach sciatic nerve block + posterior femoral cutaneous nerve block + saphenous nerve block
  Interventions: Procedure: Posterior Femoral Cutaneous Nerve Combined With Proximal Sciatic and Saphenous Nerve Block

INTERVENTIONS:
Procedure: Posterior Femoral Cutaneous Nerve Combined With Proximal Sciatic and Saphenous Nerve Block — All nerve blocks were performed under ultrasound guidance，single supragluteal approach sciatic nerve block using a nerve stimulator, 20 ml of drug was injected around the sciatic nerve, the extent of drug diffusion was observed, the needle tip was turned into the deep surface of the gluteus maximus muscle below the deep gluteal artery and 5 ml of drug was injected, followed by a retractile canal saphenous nerve block injected with 15 ml of drug, and the difference in sensation of the posterior thighs of the bilateral thighs was measured after 15 min to ensure posterior femoral cutaneous nerve were blocked
  Other Names: supragluteal approach sciatic nerve block
  Arms: Combined posterior femoral cutaneous nerve block group (Group P)
Procedure: Simple Sciatic and Saphenous Nerve Blocks — All nerve blocks were performed under ultrasound guidance，single subgluteal approach sciatic nerve block using a nerve stimulator, with 25 ml of drug injected around the sciatic nerve, followed by a retractile canal saphenous nerve block with 15 ml of drug injection
  Other Names: subgluteal approach sciatic nerve block
  Arms: Sciatic saphenous nerve block group (Group S)

SUMMARY:
The aim of this study was to observe the effects of posterior femoral cutaneous nerve block combined with sciatic and saphenous nerve block compared with sciatic and saphenous nerve block alone on postoperative posterior side of the knee (popliteal fossa) pain and sleep quality in patients with TKA, and to further alleviate postoperative posterior side of the knee pain in patients with TKA and improve the quality of postoperative sleep.

DETAILED DESCRIPTION:
Total knee arthroplasty (TKA) is one of the most common surgical procedures worldwide. Although surgical and anesthesia techniques have become more mature, poor postoperative pain control after TKA is still an important problem for patients and clinicians. Peripheral nerve blocks (PNBs) have been widely used in clinical practice for postoperative analgesia after TKA.The combinations of PNBs available for postoperative analgesia after TKA include femoral/obturator , femoral/sciatic/obturator, lumbar plexus/sciatic, and femoral/sciatic, and the combination of PNBs has been shown to be effective for postoperative analgesia after TKA in a study of TKA. Meta-analysis of postoperative pain management modalities, it was concluded that blocking multiple nerves was superior to blocking any of the nerves, periarticular infiltration, or epidural analgesia, while the combination of femoral and sciatic nerve block was overall the best postoperative analgesia for TKA. The investigators found that even in patients who underwent a single combined sciatic nerve and saphenous nerve block + continuous femoral nerve block, poor quality of sleep and pain in the affected limb were still common in the postoperative period, and the complaints of pain in the affected limb were mainly centered on the posterior side of the knee (popliteal fossa) and the margins. The area where the patient's complaints were concentrated was within the range of superficial skin sensation innervated by the posterior femoral cutaneous nerve, which is a pure sensory nerve that originates from the lumbosacral plexus, descends through the lower border of the pectineus muscle, and sends out three branches, among which the posterior femoral cutaneous branch innervates superficial sensation in the posterior thigh and popliteal fossa, and the innervation of the posterior femoral cutaneous nerve is not only limited to the posterior thigh and popliteal fossa, but may also extend to the ankle joint. even extend to the ankle joint. The investigators hypothesized that a posterior femoral cutaneous nerve block could reduce pain in the posterior side of the knee in patients after TKA, and there is a theoretically feasible anatomical basis for this hypothesis. Pain is one of the most important factors affecting the quality of sleep in patients, and pain relief may potentially improve the quality and prolong the duration of sleep in patients, thus providing the conditions for comfortable medical treatment and a good prognosis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are >45 years of age; intended to undergo elective first TKA under general anesthesia
2. ASA grade II-III.
3. Agreed to participate in this study and signed the informed consent form.
4. BMI less than 28Kg/m2.

Exclusion Criteria:

1. Patients who refuse to participate in the trial
2. Preoperative inability to communicate due to speech and hearing impairment, etc.
3. History of allergy to local anesthetics or opioids
4. Contraindications to nerve block operation.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-09-25 (Estimated); Study Completion 2024-09-25 (Estimated)

PRIMARY OUTCOMES:
Postoperative anteroposterior and posterior knee Visual Analogue Scale scores (passive motion/resting) | postoperative hour 1，postoperative hour 6，postoperative hour 24，postoperative hour 48
  The level of pain at the knee surface incision and on the posterior side of the knee at rest and motion was asked and recorded using the Visual Analogue Scale scores at postoperative hour 1 (before the patient left the PACU), postoperative hour 6, postoperative hour 24, and postoperative hour 48, respectively (0 for no pain and 10 for the most severe pain imaginable)

SECONDARY OUTCOMES:
Postoperative night sleep time | First night after surgery, second night after surgery
  Use of exercise bracelets to record actual hours of patient sleep
Earliest time on the ground | Within 48 hours of surgery
  Length of time between the end of surgery and the patient's active movement off the floor
Amount of remedial opioid use | Within 48 hours of surgery
  Total remedially applied opioids within 48 hours of surgery
Number of patient PCNA uses | Within 48 hours of surgery
  Number of times a patient presses the PCNA in the 48 hours postoperatively
Incidence rate of postoperative adverse outcomes | Within 48 hours of surgery
  Including （1）the number of people who experienced soreness in the affected limb, （2）the number of people who had nausea and the number of times they vomited,（3） the number of people who had the femoral nerve recanalized, （4）the number of people who had thrombosis in the first 48 hours after the operation, （5）and the number of people who had urinary retention.
Hip Knee Ankle | within the preoperative week versus the postoperative week
  Comparison of the change in HKA angle on lower extremity X-ray film in patients during the preoperative week versus the change in HKA angle on lower extremity X-ray film during the postoperative week

CONTACTS AND LOCATIONS:
Locations (1):
- General hospital of Ningxia medical university, Yinchuan, Ningxia, China

IPD SHARING:
Plan to Share IPD: No